CLINICAL TRIAL: NCT03510429
Title: Clinical Validation of Nutritional Supplements("Ketogenic Plus") Developed for Pancreaticobiliary Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2018-0166
Record Dates: First submitted 2018-04-17; First posted 2018-04-27 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Pancreaticobiliary Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine post-op care (Active Comparator): Routine post-op care (N=20)
  Interventions: Other: Routine post-op care
- Routine post-op care with Nutritional supplement (Experimental): Routine post-op care + Nutritional supplement by specific product (N=20)
  Interventions: Dietary Supplement: Postoperative Nutritional Supplement

INTERVENTIONS:
Dietary Supplement: Postoperative Nutritional Supplement — Postoperative Nutritional Supplement (newly developed ketogenic drink: NDKD)
  Other Names: NDKD
  Arms: Routine post-op care with Nutritional supplement
Other: Routine post-op care — Routine post-operative care
  Arms: Routine post-op care

SUMMARY:
Decreased bowel function and loss of appetite in patients who underwent pancreaticobiliary surgery contribute impaired nutritional status in postoperative period. It can also affect perioperative and oncologic outcomes negatively. Therefore it is important to improve nutritional status in postoperative period by supply tailor-made optimal diets. The investigators have developed customized postoperative diets and products for pancreaticobiliary cancer patients. This time, newly developed ketogenic drink contain beefsteak mint.

The investigators expect that nutritional supplement for pancreaticobiliary patients will increase the food intake rate and contribute a improvement of perioperative outcomes and even oncologic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age more than 19)
* Pancreaticobiliary cancer patient who is scheduled pancreaticoduodenectomy or distal pancreatectomy
* Pancreatic cancer / Duodenal cancer / Distal bile duct cancer / Ampulla of Vater cancer

Exclusion Criteria:

* Patient who denied clinical trial
* Diabetes Mellitus(DM) patient with DM complication
* Hyperlipidemia patient with vascular co-morbidity
* Impaired renal function or renal failure (GFP<70%)
* Poor nutritional status (PG-SGA grade C)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-12 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Food Intake Rate(%) for postoperative diet | 1 day before operation
  Diet Intake Rate measured by dietary satisfaction questionnaire
Food Intake Rate(%) for postoperative diet | 3 days after food intake
  Diet Intake Rate measured by dietary satisfaction questionnaire
Food Intake Rate(%) for postoperative diet | at the discharge date (8 weeks after operation)
  Diet Intake Rate measured by dietary satisfaction questionnaire
Food Intake Rate(%) for postoperative diet | at the first follow up date (4 weeks after discharge)
  Diet Intake Rate measured by dietary satisfaction questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Hepatobiliary and Pancreatic Surgery, Department of Surgery, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided